CLINICAL TRIAL: NCT06903936
Title: Comparison of the Effects of Ultrasound-guided Genicular Nerve Block and Conventional Physical Therapy on Pain, Functionality and Balance in Patients With Knee Osteoarthritis
Brief Title: Comparison of the Effect of Genicular Nerve Block and Physical Therapy in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hacer Irem Altay Caglar, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/471
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: geniculer nerve block; treatment of knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Population Groups; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: the investigator and the outcomes Assessor are different people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: GNB (GENICULAR NERVE BLOCK) group (Experimental): Group 1; GNB (GENICULAR NERVE BLOCK) group: Injection will be performed by a physiatrist with clinical experience using a linear probe with inplane technique under USG guidance.
  The patient will lie in the supine position with a pillow under the ipsilateral popliteal fossa to see the injection site easily. 6 ml of solution consisting of 5 ml 2% lidocaine hydrochloride and 1 ml 40 mg triamcinolone acetonide will be injected equally into the superomedial, inferomedial and superolateral genicular nerve branches using a 23G (0.6*60mm) needle under ultrasound guidance.
  The injector tip will be changed after each injection. Exercises will be asked to be done every day, 2 times a day, 10 repetitions for 3 weeks. The use of NSAIDs will be restricted during the treatment period.
  Interventions: Other: Group 1: GNB (GENICULAR NERVOUS NERVOUS BLOCK) group:; Other: Group 3: Exercise group
- Group 2: PT (PHYSICAL THERAPY) group: (Experimental): Group 2: PT (PHYSICAL THERAPY) group: In the PT group, all interventions will be performed with the patient supine and knees in extension. First, superficial heating will be applied using a hotpack for 20 minutes, followed by therapeutic ultrasound in continuous mode at a frequency of 1 MHz and 1.5 Watt/cm2 for 5 minutes to achieve deep thermal effects. Conventional transcutaneous electrical nerve stimulation (TENS) will then be applied for 15 minutes for a total of 15 sessions.
  Exercises will be asked to be performed 10 repetitions 2 times a day, every day for 3 weeks. NSAID use will be restricted during the treatment period.
  Interventions: Other: Group 2: PT (PHYSICAL THERAPY) group; Other: Group 3: Exercise group
- Group 3: Exercise group (Experimental): Group 3: Exercise group: For 3 weeks, exercise therapy will be applied by the patient. Knee range of motion exercises, quadriceps strengthening exercises, hamstring stretching exercises will be taught to the patients by the physician and they will be asked to perform 10 repetitions 2 times a day, every day for a total of 3 weeks. The use of NSAIDs will be restricted during the treatment period.
  The exercises will be taught to all 3 groups and they will be asked to do 10 repetitions 2 times a day, every day for 3 weeks. NSAID use will be restricted during the treatment period.
  Interventions: Other: Group 3: Exercise group

INTERVENTIONS:
Other: Group 1: GNB (GENICULAR NERVOUS NERVOUS BLOCK) group: — 6 ml of solution consisting of 5 ml 2% lidocaine hydrochloride and 1 ml 40 mg triamcinolone acetonide will be injected equally into the superomedial, inferomedial and superolateral genicular nerve branches using a 23G (0.6*60mm) needle under ultrasound guidance.
  Arms: Group 1: GNB (GENICULAR NERVE BLOCK) group
Other: Group 2: PT (PHYSICAL THERAPY) group — Group 2: PT (PHYSICAL THERAPY) group: In the PT group, all interventions will be performed with the patient supine and knees in extension. First, superficial heating will be applied using a hotpack for 20 minutes, followed by therapeutic ultrasound in continuous mode at a frequency of 1 MHz and 1.5 Watt/cm2 for 5 minutes to achieve deep thermal effects. Then traditional transcutaneous electrical nerve stimulation (TENS) will be applied for 15 minutes for a total of 15 sessions.
  Arms: Group 2: PT (PHYSICAL THERAPY) group:
Other: Group 3: Exercise group — Group 3: Control group: For 3 weeks, exercise therapy will be applied by the patient. Knee range of motion exercises, quadriceps strengthening exercises, hamstring stretching exercises will be taught to the patients by the doctor and they will be asked to do them every day, 2 times a day, 10 repetitions for a total of 3 weeks. The use of NSAIDs will be restricted during the treatment period.

SUMMARY:
Knee arthritis is a chronic joint disease that causes pain, disability and impaired quality of life, leading to significant social and health problems worldwide. Moreover, these public and economic impacts related to osteoarthritis of the knee are expected to increase in the future. With the global increase in the proportion of the elderly population, overall obesity rates and the associated incidence of osteoarthritis of the knee, clinicians are now focusing on new treatment strategies. The diagnosis is usually made by history, physical examination and radiography (X-ray) and there is no need for additional examination.

Today, both non-surgical and surgical interventions are used in the treatment of knee arthritis. Non-surgical options include patient education, weight loss, physical therapy (PT), support or foot orthosis, oral painkillers, non-cortisol anti-inflammatory drugs, cortisols, hyaluronic acid, plasma injections rich in platelets, prolotherapy, stem cell therapy and genicular nerve blocks.

The aim of the study was to compare the benefits of genicular nerve block and physical therapy in volunteers with knee pain for more than 3 months like you and to determine the most appropriate method.

In this study, Genicular nerve block and Physical therapy in patients with knee arthritis;

* Effects on knee pain, mobility and functional ability
* It is aimed to examine the effects on equilibrium parameters.

A total of 66 participants will be included in the study. Participants will be randomly assigned to three groups by envelope selection method. Your treatment method will be determined according to the treatment method in the envelope you choose.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a chronic joint disease that causes pain, disability and impaired quality of life, leading to significant social and health problems worldwide. Moreover, these public and economic impacts related to KOA are expected to increase in the future. With the global increase in the proportion of the elderly population, overall obesity rates and the associated incidence of KOA, clinicians are now focusing on new treatment strategies.

Currently, both non-surgical and surgical interventions are used to treat KOA. Non-surgical options include patient education, self-management strategies, weight loss, physical therapy (PT), brace or foot orthosis, oral analgesics, non-steroidal anti-inflammatory drugs, steroids, hyaluronic acid, platelet-rich plasma injections, prolotherapy stem cell therapy and genicular nerve blocks, all aimed at relieving pain, improving function and delaying the need for surgery. PT is an established and evidence-based treatment option for reducing pain and improving function in KOA.

Through the use of PT modalities such as thermal therapies, therapeutic ultrasound, electrical stimulation and laser therapy, which are known to modulate inflammation, are known to have an impact on pain, function and quality of life. On the other hand, genicular nerve block (GNB) is a recently developed treatment option for KOA that targets the three sensory nerves of the knee (superior lateral, superior medial and inferior medial genicular nerve) to block pain transmission to the central nervous system. Only a few studies have been conducted using GNB in patients with chronic KOA, demonstrating a reduction in pain and improvement in knee function. Eventually, GNB gained popularity in rheumatology to modulate inflammation in patients with rheumatoid arthritis. Studies investigating different methods of application of GNB in chronic KOA, namely ultrasound-guided and fluoroscopy-guided GNB, reported no difference in treatment efficacy between the two methods. However, Kim et al. reported that ultrasound is more suitable for imaging because it does not require radiation exposure.

The aim of this study was to compare the effects of genicular nerve block and physical therapy on knee pain, mobility, functional ability and balance parameters in patients with knee osteoarthritis (KOA) and to investigate whether they are superior to the control group.

ELIGIBILITY:
INCLUSION CRITERIA

* Being between forty and seventy years old
* Kellgren-Lawrence grade two-thee radiological osteoarthritis
* Knee pain for at least three months
* Those who consented to participate in the study according to the informed consent form

EXCLUSION CRITERIA

* Pregnancy
* Malignancy
* Epilepsy
* History of cardiac pacemaker
* Those who have received glucocorticosteriod, hyaluronic acid, PRP, Genicular block injection in the last six months
* Those who received physical therapy in the last six months
* Those taking oral glucosamine in the last six months
* Anticoagulant use
* History of systemic inflammatory disease
* History of fracture and surgery in the lower extremity
* Open wounds on the knees
* History of systemic infection in the patient
* Inability of the patient to cooperate
* History of neuromuscular disease affecting balance parameters
* Patient's unwillingness to participate in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | before treatment (week 0)
  Visual analog scale (VAS), pain intensity is usually graded as "no pain" 0 points and "the most severe pain imagined" 10 points (10 cm scale). Scoring intervals in pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain. VAS is a practical scale widely used in chronic pain worldwide.As the VAS score increases, the severity of pain increases.
Visual analog scale (VAS) | at the end of treatment (week 3)
  Visual analog scale (VAS), pain intensity is usually graded as "no pain" 0 points and "the most severe pain imagined" 10 points (10 cm scale). Scoring intervals in pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain. VAS is a practical scale widely used in chronic pain worldwide.As the VAS score increases, the severity of pain increases.
Visual analog scale (VAS) | 9 weeks after treatment (week 12)
  Visual analog scale (VAS), pain intensity is usually graded as "no pain" 0 points and "the most severe pain imagined" 10 points (10 cm scale). Scoring intervals in pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain. VAS is a practical scale widely used in chronic pain worldwide.As the VAS score increases, the severity of pain increases.
WOMAC index (Western Ontario and McMaster Universities to assess knee functionality) | before treatment (week 0)
  WOMAC index (Western Ontario and McMaster Universities to assess knee functionality): It consists of three subscales: Pain (5 questions), stiffness (2 questions) and function (17 questions). Total scores range from 0 to 96, with higher scores indicating poor functioning. The validity and reliability of the WOMAC index has been demonstrated in Turkish DOA patients.
WOMAC index (Western Ontario and McMaster Universities to assess knee functionality) | at the end of treatment (week 3)
  WOMAC index (Western Ontario and McMaster Universities to assess knee functionality): It consists of three subscales: Pain (5 questions), stiffness (2 questions) and function (17 questions). Total scores range from 0 to 96, with higher scores indicating poor functioning. The validity and reliability of the WOMAC index has been demonstrated in Turkish DOA patients.
WOMAC index (Western Ontario and McMaster Universities to assess knee functionality) | 9 weeks after treatment (week 12)
  WOMAC index (Western Ontario and McMaster Universities to assess knee functionality): It consists of three subscales: Pain (5 questions), stiffness (2 questions) and function (17 questions). Total scores range from 0 to 96, with higher scores indicating poor functioning. The validity and reliability of the WOMAC index has been demonstrated in Turkish DOA patients.

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | before treatment (week 0)
  6-minute walk test (6MWT): Patients would be asked to walk at their preferred pace for 6 minutes along a 30m corridor marked at 3m intervals; rest or change in walking speed would be allowed if necessary. The maximum distance covered in 6 minutes along the 30m corridor will be measured.The purpose of the 6-minute walking test is to evaluate whether patients respond to the given treatment.
6-minute walk test (6MWT) | at the end of treatment (week 3)
  6-minute walk test (6MWT): Patients would be asked to walk at their preferred pace for 6 minutes along a 30m corridor marked at 3m intervals; rest or change in walking speed would be allowed if necessary. The maximum distance covered in 6 minutes along the 30m corridor will be measured.The purpose of the 6-minute walking test is to evaluate whether patients respond to the given treatment.
6-minute walk test (6MWT) | 9 weeks after treatment (week 12)
  6-minute walk test (6MWT): Patients would be asked to walk at their preferred pace for 6 minutes along a 30m corridor marked at 3m intervals; rest or change in walking speed would be allowed if necessary. The maximum distance covered in 6 minutes along the 30m corridor will be measured.The purpose of the 6-minute walking test is to evaluate whether patients respond to the given treatment.
Notthingam activities of daily living scale | before treatment (week 0)
  Notthingam activities of daily living scale: It consists of 4 subsections; mobility (6 items), kitchen (5 items), household (5 items) and leisure activities (6 items). Responses to all questions are evaluated.
  not done, 0 points; with help, 1 point; done on own with difficulty, 2 points; done easily on own, 3 points. The total scores for each subsection and the sum of the scores for all subsections give the final total Notthingam activities of daily living scale scores ranging from 0 to 66 points.High scores indicate good performance in daily life activities.
Notthingam activities of daily living scale | at the end of treatment (week 3)
  Notthingam activities of daily living scale: It consists of 4 subsections; mobility (6 items), kitchen (5 items), household (5 items) and leisure activities (6 items). Responses to all questions are evaluated.
  not done, 0 points; with help, 1 point; done on own with difficulty, 2 points; done easily on own, 3 points. The total scores for each subsection and the sum of the scores for all subsections give the final total Notthingam activities of daily living scale scores, ranging from 0 to 66 points.High scores indicate good performance in daily life activities.
Notthingam activities of daily living scale | 9 weeks after treatment (week 12)
  Notthingam activities of daily living scale: It consists of 4 subsections; mobility (6 items), kitchen (5 items), household (5 items) and leisure activities (6 items). Responses to all questions are evaluated.
  not done, 0 points; with help, 1 point; done on own with difficulty, 2 points; done easily on own, 3 points. The total scores for each subsection and the sum of the scores for all subsections give the final total Notthingam activities of daily living scale scores, ranging from 0 to 66 points.High scores indicate good performance in daily life activities.
Measurement of Balance Parameters on the Biodex Balance Device | before treatment (week 0)
  Measurement of Balance Parameters on the Biodex Balance Device: In this study, postural stability and fall risk (total score, anteroposterior, mediolateral and overall stability) will be assessed on the Bioedex balance device before treatment (week 0), at the end of treatment (week 3) and 9 weeks after treatment (week 12).
  To avoid bias during measurements and surveys, the measurer will be blinded to the participants.
  A high score on overall balance indicates poor balance. The overall stability index is believed to be the best indicator of a patient's overall ability to balance the platform. In this study, we evaluated static balance on the Biodex balance device.
  Medio-lateral stability index (MLSI), anterior-posterior stability index (APSI), overall stability index (OSI) are standard deviations assessing fluctuations around the zero point from the horizontal rather than around the group mean. Higher values indicate more deviations and poor balance control.
Measurement of Balance Parameters on the Biodex Balance Device | at the end of treatment (week 3)
  Measurement of Balance Parameters on the Biodex Balance Device: In this study, postural stability and fall risk (total score, anteroposterior, mediolateral and overall stability) will be assessed on the Bioedex balance device before treatment (week 0), at the end of treatment (week 3) and 9 weeks after treatment (week 12).
  To avoid bias during measurements and surveys, the measurer will be blinded to the participants.
  A high score on overall balance indicates poor balance. The overall stability index is believed to be the best indicator of a patient's overall ability to balance the platform. In this study, we evaluated static balance on the Biodex balance device.
  Medio-lateral stability index (MLSI), anterior-posterior stability index (APSI), overall stability index (OSI) are standard deviations assessing fluctuations around the zero point from the horizontal rather than around the group mean. Higher values indicate more deviations and poor balance control.
Measurement of Balance Parameters on the Biodex Balance Device | 9 weeks after treatment (week 12)
  Measurement of Balance Parameters on the Biodex Balance Device: In this study, postural stability and fall risk (total score, anteroposterior, mediolateral and overall stability) will be assessed on the Bioedex balance device before treatment (week 0), at the end of treatment (week 3) and 9 weeks after treatment (week 12).
  To avoid bias during measurements and surveys, the measurer will be blinded to the participants.
  A high score on overall balance indicates poor balance. The overall stability index is believed to be the best indicator of a patient's overall ability to balance the platform. In this study, we evaluated static balance on the Biodex balance device.
  Medio-lateral stability index (MLSI), anterior-posterior stability index (APSI), overall stability index (OSI) are standard deviations assessing fluctuations around the zero point from the horizontal rather than around the group mean. Higher values indicate more deviations and poor balance control.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer I Altay Caglar, ra, Principal Investigator — Kirsehir Ahi Evran University Physical Medicine and Rehabilitation Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Kirsehir Ahi Evran University Physical Medicine and Rehabilitation Hospital, Kirşehi̇r, Kirşehi̇r
  - Ahi Evran University Hospital, Kırşehir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sert AT, Sen EI, Esmaeilzadeh S, Ozcan E. The Effects of Dextrose Prolotherapy in Symptomatic Knee Osteoarthritis: A Randomized Controlled Study. J Altern Complement Med. 2020 May;26(5):409-417. doi: 10.1089/acm.2019.0335. Epub 2020 Mar 30. PMID 32223554
- [Background] Kim DH, Lee MS, Lee S, Yoon SH, Shin JW, Choi SS. A Prospective Randomized Comparison of the Efficacy of Ultrasound- vs Fluoroscopy-Guided Genicular Nerve Block for Chronic Knee Osteoarthritis. Pain Physician. 2019 Mar;22(2):139-146. PMID 30921977
- [Background] Fu Y, Du Y, Li J, Xi Y, Ji W, Li T. Demonstrating the effectiveness of intra-articular prolotherapy combined with peri-articular perineural injection in knee osteoarthritis: a randomized controlled trial. J Orthop Surg Res. 2024 May 5;19(1):279. doi: 10.1186/s13018-024-04762-4. PMID 38705988